CLINICAL TRIAL: NCT02057120
Title: INFLUENCE OF KINESIO TAPING ON MUSCLE ACTIVATION, MUSCLE STRENGTH AND PERFORMANCE JUMP IN YOUNG ATHLETES. CLINICAL STUDY, RANDOMIZED, PLACEBO-CONTROLLED AND DOUBLE BLIND
Brief Title: Influence of Kinesio Taping on Muscle Activation, Muscle Strength and Performance of Young Football Athletes Jump
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Doctor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21892213.4.0000.5511
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-12

CONDITIONS: Kinesio Taping
Keywords: Kinesio Taping, Soccer, Hop Test, Electromyography, Athletic Performance, Muscle Strength Dynamometer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Grupo A (Kinesio Taping) (Active Comparator): Will be held the application of Kinesio Taping (Tex Gold) in the region of the rectus femoris dominant lower limb by a physical therapist trained in the technique (KT1 KT2 and) and with experience in this type of application to be designed without knowing in which group fits this patient. In the sequence, the athlete will be oriented to remain at rest for 30 min to get a better grip on the tape and one of the first tests and rest, only after this period will conduct a new evaluation of jump tests (single leg Hop test and Triple Hop Test) and, finally, a new test of strength in the isokinetic dinamomêtro in conjunction with the electromyographic assessment.
  Interventions: Procedure: Kinesio Taping
- Placebo Taping (Placebo Comparator): The volunteer will receive a Placebo application tape, being in this case the physical therapist will apply a strip of Kinesio Taping perpendicular to the muscle fibers of the rectus femoris of the dominant member of the individual.
  Interventions: Device: Kinesio Taping placebo

INTERVENTIONS:
Procedure: Kinesio Taping — Application of Kinesio (Kinesio Tex Gold ®) of black color. The tape will be applied from proximal to distal, leaving the anterosuperior iliac spine Bottom, passing over the Rectus Femoris and ending in the region of the anterior tibia tuberosity with a voltage of 25 %.
  Arms: Grupo A (Kinesio Taping)
Device: Kinesio Taping placebo — The volunteer who is allocated at random in the placebo group will receive an application of Kinesio transverse way the rectus femoris muscle, in order to verify a possible placebo effect of application of tape.
  Arms: Placebo Taping

SUMMARY:
The objective of the project is to investigate the influence of application of Kinesio Taping in young athletes in football, muscle strength and muscle activation in the performance of the Single Leg Hop Test tests and Triple Hop Test methods: will be conducted a randomized, placebo-controlled and double-blind. 24 individuals will be athletes who fit the criteria for inclusion will be randomized into 2 groups (Placebo, Kinesio Taping Taping) and will be submitted to the tests of Single Leg Hop Test, Triple Hop Test, the isokinetic evaluation and electromyographic of Rectus Femoris dominant lower limb. Then the intervention shall be carried out with application of Kinesio Taping for activation of rectus femoris muscle group and placebo intervention Kinesio Taping with application of Kinesio Taping of transverse way the rectus femoris without tension in the Placebo group Taping. The volunteers will be re-evaluated 30 minutes after application of the technique and 12:0 am after with the same tests for that later can be compared the results obtained in each group. Analysis: will be achieved statistical tests and adopted a significance level of 5 percent

DETAILED DESCRIPTION:
The method of bandage with Kinesio Taping created by Kenzo Kase in 1996, it is the application of a thin, elastic tape with a thickness similar to the epidermis, on the skin. Being that it can be stretched up to 140 of its original length making it elastic enough compared to the conventional bandages. Kenzo still claims that the tape is able to reduce pain, swelling, muscle spasms and prevent injury. As much as there is today a widespread use of this technique mainly in the context of sports and orthopedics, still lack reliable studies to support the theory described by this method. Objectives: to investigate the influence of application of Kinesio Taping in young athletes in football, muscle strength and muscle activation in the performance of the Single Leg Hop Test tests and Triple Hop Test methods: will be conducted a randomized, placebo-controlled and double-blind. 24 individuals will be athletes who fit the criteria for inclusion will be randomized into 2 groups (Placebo, Kinesio Taping Taping) and will be submitted to the tests of Single Leg Hop Test, Triple Hop Test, the isokinetic evaluation and electromyographic of Rectus Femoris dominant lower limb. Then the intervention shall be carried out with application of Kinesio Taping for activation of rectus femoris muscle group and placebo intervention Kinesio Taping with application of Kinesio Taping of transverse way the rectus femoris without tension in the Placebo group Taping. The volunteers will be re-evaluated 30 minutes after application of the technique and 12:0 am after with the same tests for that later can be compared the results obtained in each group. Analysis: will be achieved statistical tests and adopted a significance level of 5 percent.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 15 and 20 years, Football players and Athletes who have body mass index (BMI) considered normal (between 20 and 25).

Exclusion Criteria:

* History of lower limb musculoskeletal injuries in the last 6 months, history of lower limb and spine surgery in the last 6 months and BMI over 25 or less than 20.

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hop Test | 1 year
  The volunteer must position themselves in foot with unipodal support in the dominant lower limb behind a line that will be demarcated on the ground and jump as far as possible, without support in the contralateral limb or imbalance. The distance will be measured with a tape measure, from the starting point (line demarcated on the ground) until the most proximal point of the heel of the foot fell on the floor.

SECONDARY OUTCOMES:
Surface electromyography | 1 year
  During isokinetic evaluation will also be carried out a study of the electrical activity of the rectus femoris muscle. For the capture of the electrical signal of that muscle will be used the acquisition system with 8 channels (EMG System of Brazil Ltda ®), composed of active electrodes with bipolar won 20 times amplification, analog filter pass band of 20 to 500 Hz and common mode rejection of 120 dB, and one of the channels will be enabled to use the force transducer (EMG System of Brazil Ltda ®). EMG signals are sampled with 2000 Hz frequency, scanned for AD conversion plate (analog-digital) with 16 bits of resolution.

OTHER OUTCOMES:
Isokinetic evaluation of knee Extensors | 1 year
  Immediately after heating and evaluation of jumps, the volunteers will perform the test of maximum voluntary contraction (CVM). Being they, positioned sitting on the seat of the isokinetic dynamometer (4, Biodex) the dominant limb is positioned to 60° of knee flexion (with 0° corresponds to total knee extension) and attached to the seat by means of a dynamometer belt. The non-dominant lower limb will also be positioned with 100° of flexion of hip and will also be attached to the seat with a belt. The volunteers will also be attached to the seat of the dynamometer through two belts across his torso. During the tests the volunteers will be instructed to place his arms across the trunk and the dynamometer axis is positioned parallel to the center of the knee joint. The CVM test will consist in the execution of three isometric contractions of knee extensors of the non-dominant lower limb with duration of 5 seconds, the highest torque value obtained in the three contractions (peak torque).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: URL of the University of Nove de Julho — http://www.uninove.br